CLINICAL TRIAL: NCT03781336
Title: Brief Mindfulness Meditation Course to Reduce Stress in Healthcare Professionals and Trainees: A Randomized Clinical Trial
Brief Title: Brief Mindfulness Meditation Course to Reduce Stress in Healthcare Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Rezvan Ameli, Principal Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-MH-0018
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Stress, Professional; Stress, Psychological
Keywords: mindfulness; stress; resilience building; meditation; healthcare professionals; trainees; physicians; nurses
MeSH Terms: conditions — Occupational Stress; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants are allocated into the mindfulness-based self-care group or a wait list group for 5 weeks. Since the group is offered during work hours, the waitlist group could be best described as "life as usual". After group allocation, all participants completed demographic and self report clinical assessments at baseline, and self report clinical assessments at follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based self-care (Experimental): Mindfulness-based self-care (5 weeks)
  Interventions: Behavioral: Mindfulness-based self care
- Life as usual control (No Intervention): Life as usual control (5 weeks)

INTERVENTIONS:
Behavioral: Mindfulness-based self care — Experimental: an abridged mindfulness-based program that is incorporated into the work day, which consists of five weekly 1.5 hour sessions.
  Arms: Mindfulness-based self-care

SUMMARY:
Stress among healthcare professionals is well documented. Untreated stress can lead to anxiety, depression, substance use, and suicide. The use of mindfulness-based programs to reduce stress and enhance wellbeing, among health care professionals, has increased with promising results. Typical mindfulness-based programs are 30 hours in length across 9 sessions. The purpose of this study is to assess the effectiveness of a shorter and more practical program that could be offered during work hours to health care professionals at the NIH Clinical Center. The program will be delivered in five weekly 1.5 hour sessions.

DETAILED DESCRIPTION:
This abridged program was designed by Dr. Rezvan Ameli who is an expert in mindfulness-based practices/therapies and was in response to the expressed needs of the NIH clinical staff and the NIH fellowship training program.

Participants completed all primary and secondary outcome measure questionnaires at week -1, 5 and 13. The life as usual control group completed all primary and secondary outcome measures at week -1, and 5.

The program is described below:

The program consisted of 5 sessions. A class binder was prepared for the participants and included information about mindfulness and its practice, practices covered in each session, Practice Plan work sheets to design home practices, pertinent reference list, guide to online services, programs and apps, selected poetry, and information regarding recorded instructions for body scan and mindful breathing by the instructor which was made available on the institution's website and could be downloaded by the participants. Each session was 1.5 hours in length and was offered on Fridays from 3-4:30 pm. Classes were instructed by Rezvan Ameli, Ph.D., clinical psychologist, an experienced mindfulness practitioner since 2003 and teacher since 2008. In addition to her background as a licensed clinical psychologist, mindfulness practitioner, teacher and writer (Ameli 2013), RA is a certified yoga teacher and is registered with the Yoga Alliance (RYT-200).

Common Elements of the Sessions

The first 4 classes began with 20-25 minutes of mindful movement/ light yoga (TNH sounds true, ITP kata). We did not include movements in the 5th (last) session due to time constraints. The emphasis during mindful movements was on the coordination of movement and the breath with the instruction that when the mind wandered away to gently bring it back and refocus on the breath and movements. Participants were encouraged to only engage in movements that felt comfortable but not straining, painful, or felt unsafe. Each class had a period of "check in". During the first check in, participants shared their names, a brief statement about the reason for their participation, and their current self-care practice/s if any. Class guidelines including confidentiality were reviewed at this time. In subsequent check-ins the participants addressed their questions regarding mindfulness practices and class teachings, described their practice with a focus on self-care, their existing self-care practices and new learnings from the class, and any obstacles to their practice and to their self-care during the preceding week. Other common elements of the sessions included a period of inquiry, i.e. question and answer, after each new practice was introduced, planning a week of practice based on class learnings, post class ratings, and concluding the class with a relevant poem. Home practice planning was done in dyads of participants who were then encouraged to stay in touch, become a "buddy" to their class partner, and communicate during the week about their practice. Every session included a period of mindful breathing. The length of mindful breathing (sitting meditation) was gradually increased from 10 minutes in the 1st session to 30 minutes in the 5th session.

Session Specific Practices

In addition to these common elements, each session included a theme and other specific mindfulness practices as follows:

* Session 1- Theme: Introduction to mindfulness. This session included definition of mindfulness and its foundations (Kabat-Zin, 1992), mindful breathing and body scan.
* Session 2- Theme: Enhancing Awareness & Focused Attention. This session included mindfulness of sounds, a short body scan, mindful breathing, and mindful eating, i.e. the "raisin exercise" (ref). In addition, a discussion of mindful consumption and its relevance to self-care was explored (Ameli 2013).
* Session 3 -Theme: Awareness of pleasurable experiences. This session included mindfulness of the breath (briefly incorporating sounds, body sensation, thoughts, feelings and then focusing on the breath), and mindful walking. The importance of awareness of pleasurable experiences were discussed and an exercise to enhance attention to pleasurable experiences was performed in dyads (Ameli 2013).
* Session 4- Theme: Transformation of difficult emotions through mindfulness. In this session the concept of transforming difficult emotions through the practice of mindfulness was discussed, explored, and practiced. The acronym RAIN (recognize, accept/allow, investigate, and non-identification) was utilized to facilitate this practice.
* Session 5- Theme: Compassion. This session mindful breathing and a general discussion of compassion, compassion towards self and other, and the practice of loving kindness (Ameli 2013). The class was concluded with a "check-out" where participants briefly shared their overall experiences and learnings and their goals/vision for future self-care activities and practices.

ELIGIBILITY:
Inclusion Criteria:

* Any National Institutes of Health (NIH) employee, contractor, or trainee willing and able to participate in a 5-week mindfulness-based self-care course during the work day.
* English speaking

Exclusion Criteria

* Persons with medical and psychiatric conditions were advised to consult with their health care practitioners prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rezvan Ameli, PhD, Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ameli, R. (2013). 25 Lessons in Mindfulness : Now Time for Healthy Living (First edition. ed.). Washington, D.C.: American Psychological Association.
- [Background] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563
- [Background] de Vibe M, Solhaug I, Rosenvinge JH, Tyssen R, Hanley A, Garland E. Six-year positive effects of a mindfulness-based intervention on mindfulness, coping and well-being in medical and psychology students; Results from a randomized controlled trial. PLoS One. 2018 Apr 24;13(4):e0196053. doi: 10.1371/journal.pone.0196053. eCollection 2018. PMID 29689081
- [Background] West CP, Dyrbye LN, Erwin PJ, Shanafelt TD. Interventions to prevent and reduce physician burnout: a systematic review and meta-analysis. Lancet. 2016 Nov 5;388(10057):2272-2281. doi: 10.1016/S0140-6736(16)31279-X. Epub 2016 Sep 28. PMID 27692469
- [Background] Dyrbye LN, Shanafelt TD. Physician burnout: a potential threat to successful health care reform. JAMA. 2011 May 18;305(19):2009-10. doi: 10.1001/jama.2011.652. No abstract available. PMID 21586718
- [Background] West CP, Dyrbye LN, Rabatin JT, Call TG, Davidson JH, Multari A, Romanski SA, Hellyer JM, Sloan JA, Shanafelt TD. Intervention to promote physician well-being, job satisfaction, and professionalism: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):527-33. doi: 10.1001/jamainternmed.2013.14387. PMID 24515493
- [Derived] Ameli R, Sinaii N, West CP, Luna MJ, Panahi S, Zoosman M, Rusch HL, Berger A. Effect of a Brief Mindfulness-Based Program on Stress in Health Care Professionals at a US Biomedical Research Hospital: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2013424. doi: 10.1001/jamanetworkopen.2020.13424. PMID 32840621
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Started | 45 | 37
Completed | 43 (All participants were included in the analysis (Intent to treat)) | 35 (All participants were included in the analysis (Intent to treat))
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-based Self-care | Life as Usual Control | Total
Number analyzed (Participants) | 43 | 35 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (15.4) | 36.4 (13.0) | 36.0 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 28 | 65
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 38 | 30 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 27 | 21 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Marital status [Count of Participants; unit: Participants]
  Single | 28 | 19 | 47
  Married | 8 | 12 | 20
  Divorced or separated | 3 | 3 | 6
  Widowed or other | 4 | 1 | 5
Religion [Count of Participants; unit: Participants]
  Agnostic | 1 | 2 | 3
  Atheism | 5 | 3 | 8
  Buddhism | 2 | 2 | 4
  Christianity | 18 | 13 | 31
  Hinduism | 3 | 2 | 5
  Islam | 2 | 3 | 5
  Judaism | 2 | 2 | 4
  Not affiliated or other | 10 | 8 | 18
Current position [Count of Participants; unit: Participants]
  Administrator | 7 | 3 | 10
  Nurse | 2 | 3 | 5
  PhD Scientist | 6 | 3 | 9
  Physician | 7 | 11 | 18
  Social Worker | 2 | 3 | 5
  Training Fellow | 19 | 12 | 31
Education level [Count of Participants; unit: Participants]
  Some college | 1 | 1 | 2
  Completed college | 22 | 14 | 36
  Graduate school or Advance degree | 20 | 20 | 40
Preexisting condition [Number; unit: participants]
  Medical condition | 16 | 9 | 25
  Psychiatric condition | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale (PSS) is used to assess self-reported perceived stress. It is a 10-item scale, with a total range from 0 (no symptoms) to 40 (highest severity).
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
score on a scale
  Baseline | 19.63 (6.26) | 18.80 (6.36)
  Postintervention | 17.29 (5.84) | 18.54 (6.30)
  Follow-up | 13.80 (6.45) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

2. Secondary Outcome: Mindful Attention Awareness Scale (MAAS) - Trait Version
Description: The Mindful Attention Awareness Scale-Trait Version (MAAS-T) is used to assess self-reported trait mindfulness. It is a 15-item scale, with a total range from 0 (low mindfulness) to 90 (high mindfulness).
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
score on a scale
  Baseline | 3.74 (0.99) | 3.61 (0.89)
  Postintervention | 3.95 (0.83) | 3.70 (0.96)
  Follow-up | 4.33 (0.85) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

3. Secondary Outcome: Mindful Attention Awareness Scale (MAAS) - State Version
Description: The Mindful Attention Awareness Scale-State Version (MAAS-S) is used to assess self-reported state mindfulness. It is a 5-item scale, with a total range from 0 (high mindfulness) to 30 (low mindfulness).
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
score on a scale
  Baseline | 2.23 (1.24) | 2.48 (1.08)
  Postintervention | 3.74 (1.18) | 2.78 (1.16)
  Follow-up | 4.08 (1.04) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

4. Secondary Outcome: Positive Affect Scores (PANAS)
Description: The Positive And Negative Affect Scale (PANAS) is used to assess self-reported positive and negative affect. It is a two dimension scale, with total ranges for each scale from 0 (low positive/negative affect) to 50 (high positive/negative affect).
  These are the Positive Affect Scores
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
units on a scale
  Baseline | 32.85 (7.73) | 33.67 (5.95)
  Postintervention | 35.69 (7.12) | 31.42 (7.27)
  Follow-up | 36.13 (8.43) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

5. Secondary Outcome: Visual Analog Scale-Anxiety (VAS-A)
Description: Visual Analog Scale-Anxiety (VAS-A) is used to assess self-reported anxiety. It is a 1-item scale, with a total range from 1 (low anxiety) to 10 (high anxiety).
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
score on a scale
  Baseline | 4.72 (1.62) | 4.57 (1.69)
  Postintervention | 2.58 (1.52) | 4.23 (1.73)
  Follow-up | 3.29 (1.47) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

6. Secondary Outcome: Mindful Self Care Scale-General (MSCS-G)
Description: Mindful Self Care Scale-General (MSCS-G) is used to assess self-reported mindful self care. It is a 3-item scale, with a total range from 0 (low self care) to 12 (high self care).
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
score on a scale
  Baseline | 5.60 (2.75) | 6.00 (2.88)
  Postintervention | 7.29 (2.44) | 5.54 (2.77)
  Follow-up | 6.37 (2.76) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

7. Secondary Outcome: Maslach Burnout Inventory (MBI)
Description: The Maslach Burnout Inventory (MBI 2-Item) is used to assess self-reported burnout. The 2-Item inventory assesses emotional exhaustion (Item-1) and depersonalization (Item-2) separately from 1 (no symptoms) to 7 (highest severity).
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
score on a scale
  Baseline-item 1 | 2.95 (1.56) | 3.29 (1.45)
  Postintervention-item 1 | 2.89 (1.63) | 2.74 (1.62)
  Follow-up-item 1 | 2.31 (1.64) | NA (NA) — Follow-up data not collected from the life as usual control subjects.
  Baseline-item 2 | 1.76 (1.32) | 1.6 (1.42)
  Postintervention-item 2 | 1.22 (1.13) | 1.57 (1.36)
  Follow-up-item 2 | 1.34 (1.21) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

8. Secondary Outcome: Negative Affect Scores (PANAS)
Description: The Positive And Negative Affect Scale (PANAS) is used to assess self-reported positive and negative affect. It is a two dimension scale, with total ranges for each scale from 0 (low positive/negative affect) to 50 (high positive/negative affect).
  These are the Negative Affect Scores
Time Frame: Week-1(baseline), Week-5 (post-intervention), Week-13 (follow-up)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
Number analyzed (Participants) | 43 | 35
units on a scale
  Baseline | 21.44 (7.38) | 21.21 (7.27)
  Postintervention | 20.73 (6.24) | 19.09 (7.60)
  Follow-up | 18.22 (6.01) | NA (NA) — Follow-up data not collected from the life as usual control subjects.

ADVERSE EVENTS:
Time Frame: Week-5 (post-intervention)
Description: Adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov.
Arm/Group | Mindfulness-based Self-care | Life as Usual Control
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/35
Other Adverse Events (participants affected / at risk) | 0/43 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03781336/Prot_SAP_000.pdf